CLINICAL TRIAL: NCT01758523
Title: Dutasteride Treatment for the Reduction of Heavy Drinking
Brief Title: Dutasteride Treatment for the Reduction of Heavy Drinking in Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonathan Covault, Professor of Psychiatry, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-056-2; 2P60AA003510 (NIH)
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Alcoholism; Alcohol Abuse; Alcohol Dependence
Keywords: neuroactive steroids
MeSH Terms: conditions — Alcoholism | interventions — Dutasteride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dutasteride (Experimental): 4 mg oral loading dose of dutasteride followed by 1 mg/day dutasteride for 12 weeks.
  Interventions: Drug: Dutasteride
- Sugar Pill (Placebo Comparator): Placebo pills prepared to appear the same as active medication and taken in the same number as active medication for 12 weeks.
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Dutasteride
  Other Names: Avodart
  Arms: dutasteride
Drug: sugar pill
  Other Names: placebo
  Arms: Sugar Pill

SUMMARY:
This study will examine the safety and potential benefit of the medication dutasteride to help men reduce or stop drinking alcohol.

DETAILED DESCRIPTION:
Extensive preclinical studies indicate that neuroactive steroids medicate important effects of alcohol and support the examination of neuroactive steroid modulators as treatment options for alcohol use problems. Dutasteride, a widely prescribed medication for benign prostatic hypertrophy, blocks a key step in the production of neuroactive steroids and represents a promising candidate for treatment of alcohol use disorders. This study will use a 12-week randomized placebo controlled design to examine the safety and efficacy of dutasteride to reduce drinking among a sample of 160 men with hazardous levels of alcohol use. It will additionally examine the potential moderation of dutasteride treatment effects by a common missense polymorphism in a neuroactive steroid biosynthetic enzyme that we have previously reported to be associated with alcohol dependence. Identification of genetic predictors of medication response offers the potential for matching alcohol treatment medications with those most likely to respond.

ELIGIBILITY:
Inclusion Criteria:

* an average weekly ethanol consumption of at least 24 standard drinks;
* be able to read English at the 8th grade or higher level;
* no evidence of significant cognitive impairment;
* be willing to provide signed, informed consent to participate in the study (including a willingness to stop or reduce drinking to non-hazardous levels);
* be willing to nominate an individual who will know the patient's whereabouts to facilitate follow up during the study

Exclusion Criteria:

* history of significant alcohol withdrawal symptoms (e.g. substantial tremor, autonomic changes, perceptual distortions, seizures, delirium, or hallucinations);
* current Diagnostic and Statistical Manual Version IV (DSM-IV) diagnosis of Alcohol Dependence who on clinical examination by a physician, are deemed to be too severely alcohol dependent to permit them to participate in a placebo-controlled study (e.g. evidence of serious adverse medical or psychiatric effects that are exacerbated by heavy drinking and would, for safety reasons, lead the physician to urge the patient to be totally abstinent and engage in an empirically supported treatment).
* current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation,(we will not exclude patients with hypertension, diabetes mellitus, asthma or other common medical conditions, if these are adequately controlled and the patient has an ongoing relationship with a primary care provider)
* serious psychiatric illness on the basis of history or psychiatric examination (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, organic mental disorder, current clinically significant eating disorder, or substantial suicide or violence risk);
* current DSM-IV diagnosis of drug dependence (other than nicotine dependence);
* currently taking psychotropics other than medication for depression/anxiety disorder (with stable dose for at least 4 weeks),medications for treatment of Attention Deficit/Hyperactivity Disorder (with stable dose for at least 4 weeks), a non-benzodiazepine sleep medication or a low dose of benzodiazepine equivalent to 2 mg clonazepam or lorazepam per day;
* are considered by the investigators to be an unsuitable candidate for receipt of an investigational drug

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2013-01; Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Covault, M.D., PhD., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Covault J, Tennen H, Feinn R. Randomized Placebo-Controlled Clinical Trial of Dutasteride for Reducing Heavy Drinking in Men. J Clin Psychopharmacol. 2024 May-Jun 01;44(3):223-231. doi: 10.1097/JCP.0000000000001849. PMID 38684046

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 47 subjects not randomized: 23 excluded at in person screening visit; 24 subjects withdrew prior to randomization
Groups:
- Dutasteride: 4 mg oral loading dose of dutasteride followed by 1 mg/day dutasteride for 12 weeks.
  Dutasteride
- Sugar Pill: Placebo pills prepared to appear the same as active medication and taken in the same number as active medication for 12 weeks.
  sugar pill
Period: Overall Study
Arm/Group | Dutasteride | Sugar Pill
Started | 74 | 68
Attended >/= 1 Visit Post-randomization | 68 | 67
Completed | 53 | 54
Not Completed | 21 | 14
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 4 | 2
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 12 | 7

BASELINE CHARACTERISTICS:
Population: Subjects who completed at least 1 visit post-randomization (modified intention to treat sample)
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride | Sugar Pill | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 62 | 126
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (7.9) | 53.1 (9.4) | 53.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 68 | 67 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 67 | 67 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 66 | 65 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 68 | 67 | 135
Heavy Drinking Days (HDD)/wk [Mean (Standard Deviation); unit: heavy drinking days / week] — days/week with 5 or more drinks over the 60 days prior to screening visit
  heavy drinking days / week | 5.2 (2.2) | 5.2 (2.1) | 5.2 (2.1)
Drinks/week [Mean (Standard Deviation); unit: drinks/week] — Total standard drinks / week over 60 day prior to screening visit
  drinks/week | 48.8 (24) | 47.3 (20.4) | 48.0 (22.2)
AbstinentDays/week [Mean (Standard Deviation); unit: days] — Days per week with no drinking during the 60 days prior to screening visit
  days | 0.67 (1.1) | 0.62 (1.1) | 0.64 (1.1)
DSM-IV Alcohol Dependence criteria [Mean (Standard Deviation); unit: units on a scale] — Number of current Diagnostic and Statistical Manual (DSM-IV) criteria for alcohol dependence (0-7; higher number greater severity of dependence; >2 criteria required for diagnosis of alcohol dependence)
  units on a scale | 4.3 (1.6) | 4.0 (1.6) | 4.2 (1.6)
Short Inventory of Problems [Mean (Standard Deviation); unit: units on a scale] — The Short Inventory of Problems (SIP). The SIP, is a 15-item instrument with a total score that ranges from 0 to 45, higher score worse outcomes.
  units on a scale | 17.2 (8.2) | 16.8 (8.8) | 17.0 (8.4)
Smoker [Count of Participants; unit: Participants] — 5 or more cigarettes per day
  Participants | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Heavy Drinking Days Per Week
Description: Number of days / study week with 5 or more drinks consumed
Time Frame: 12-week treatment period
Population: Modified Intention to Treat (ITT) all subjects who attended one or more post-randomization visit.
Measure: Mean (Standard Error); unit: heavy drinking days/week
Arm/Group | Dutasteride | Sugar Pill
Number analyzed (Participants) | 68 | 67
heavy drinking days/week | 1.75 (0.33) | 2.67 (0.34)
Statistical Analysis 1: Comparison: Dutasteride vs Sugar Pill; Test type: Other; p = 0.002, Mixed Models Analysis

2. Primary Outcome: Drinks Per Week
Description: Total number of drinks aggregated by week
Time Frame: 12-week treatment period
Population: Modified ITT (all subjects who attended one or more post-randomization visit)
Measure: Mean (Standard Error); unit: drinks/week
Arm/Group | Dutasteride | Sugar Pill
Number analyzed (Participants) | 68 | 67
drinks/week | 22.0 (2.6) | 27.2 (2.4)
Statistical Analysis 1: Comparison: Dutasteride vs Sugar Pill; Test type: Other; p = 0.028, Mixed Models Analysis

3. Primary Outcome: Number of Participants With no Heavy Drinking Days
Description: Number of participants with no heavy drinking days (days with 5 or more drinks) during the last 4 weeks of treatment.
Time Frame: Last 4 weeks of treatment
Population: Per protocol 12-week completer
Measure: Count of Participants; unit: Participants
Arm/Group | Dutasteride | Sugar Pill
Number analyzed (Participants) | 53 | 54
Participants | 16 | 8
Statistical Analysis 1: Comparison: Dutasteride vs Sugar Pill; Test type: Other; p = 0.057, Chi-squared; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.96 to 6.45]

4. Primary Outcome: Number of Participants With no Hazardous Drinking
Description: Number of participants with no hazardous drinking (not more than 4 drinks on one day and not more than 14 drinks per week) during the last 4 weeks of treatment.
Time Frame: Last 4 weeks of treatment
Population: Per protocol 12 week treatment completers
Measure: Count of Participants; unit: Participants
Arm/Group | Dutasteride | Sugar Pill
Number analyzed (Participants) | 53 | 54
Participants | 13 | 3
Statistical Analysis 1: Comparison: Dutasteride vs Sugar Pill; Test type: Other; p = 0.007, Fisher Exact; Odds Ratio (OR) = 5.5, 95% CI 2-sided [1.5 to 20.7]

5. Secondary Outcome: HDD/ Week by Treatment Group and AKR1C3*2 Genotype
Description: Change in Number of days / week with 5 or more drinks consumed contrasting AKR1C3*2 CC vs. G-carrier genotype and treatment group
Time Frame: 12-week treatment period
Population: Modified ITT (all subjects who attended one or more post-randomization visit)
Measure: Mean (Standard Error); unit: heavy drinking days/week
Groups:
- Dutasteride - AKR1C3*2 CC: dutasteride treated AKR1C3*2 CC genotype subjects
- Sugar Pill - AKR1C3*2 CC: placebo treated AKR1C3*2 CC genotype subjects
- Dutasteride - AKR1C3*2 G-carrier: dutasteride treated AKR1C3*2 G-carrier genotype subjects
- Sugar Pill - AKR1C3*2 G-carrier: placebo treated AKR1C3*2 G-carrier genotype subjects
Arm/Group | Dutasteride - AKR1C3*2 CC | Sugar Pill - AKR1C3*2 CC | Dutasteride - AKR1C3*2 G-carrier | Sugar Pill - AKR1C3*2 G-carrier
Number analyzed (Participants) | 19 | 25 | 49 | 42
heavy drinking days/week | 1.06 (0.48) | 2.9 (0.53) | 2.05 (0.42) | 2.5 (0.44)
Statistical Analysis 1: Comparison: Dutasteride - AKR1C3*2 CC vs Sugar Pill - AKR1C3*2 CC vs Dutasteride - AKR1C3*2 G-carrier vs Sugar Pill - AKR1C3*2 G-carrier; Test type: Other; p = 0.87, Mixed Models Analysis — significance for drug x AKR1C3*2 G-carrier genotype

6. Secondary Outcome: Carbohydrate-deficient Transferrin
Description: Carbohydrate-deficient transferrin (CDT) at end of treatment as percentage of baseline. Serum CDT is a biochemical measure of heavy alcohol use.
Time Frame: end of 12-week treatment vs. baseline
Population: Per protocol 12-week completers (serum sample not available for 1 placebo subject).
Measure: Mean (Standard Error); unit: percentage of baseline CDT
Arm/Group | Dutasteride | Sugar Pill
Number analyzed (Participants) | 53 | 53
percentage of baseline CDT | 94 (3.8) | 107 (4.0)
Statistical Analysis 1: Comparison: Dutasteride vs Sugar Pill; Test type: Other; p = 0.030, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Bi-weekly during 12-week active treatment then bi-monthly for 6 months
Description: At each patient visit the study nurse used a 16-item adverse events questionnaire to screen for presence of adverse events.
Arm/Group | Dutasteride | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/67
Serious Adverse Events (participants affected / at risk) | 4/68 | 2/67
Other Adverse Events (participants affected / at risk) | 37/68 | 27/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride (N=68) | Sugar Pill (N=67)
alcohol withdrawal (Nervous system disorders) | 2 | 1
Tonsillar abscess (Infections and infestations) | 1 | 0
Chronic back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride (N=68) | Sugar Pill (N=67)
Stomach discomfort (Gastrointestinal disorders) | 11 | 3
Muscle or joint pain (Musculoskeletal and connective tissue disorders) | 11 | 7
Headache (General disorders) | 10 | 11
Reduced Libido (Reproductive system and breast disorders) | 6 | 0
Fatigue (General disorders) | 5 | 7
Sleep disturbance (General disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 4 | 5
Impotence (Reproductive system and breast disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT01758523/Prot_SAP_000.pdf